CLINICAL TRIAL: NCT06294912
Title: A Controlled Human Malaria Infection Study to Evaluate the Antimalarial Activity of MK-7602 Against Plasmodium Falciparum Blood Stage Infection in Healthy Adult Participants
Brief Title: A Study to Evaluate Antimalarial Activity and Safety of MK-7602 in Healthy Adults (MK-7602-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7602-003; MK-7602-003 (Other: MSD)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Primaquine; Artesunate; atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Panel A: MK-7602 Single dose Part 1 (Experimental): Participants are inoculated with Plasmodium falciparum (P. falciparum). Panel A participants receive MK-7602 as a single oral dose. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel B: MK-7602 Single dose Part 1 (Experimental): Participants are inoculated with P. falciparum. Panel B participants receive MK-7602 as a single oral dose. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel C: MK-7602 Single dose Part 1 (Experimental): Participants are inoculated with P. falciparum. Panel C participants receive MK-7602 as a single oral dose. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel D: MK-7602 Single dose Part 1 (Experimental): Participants are inoculated with P. falciparum. Panel D participants receive MK-7602 as a single oral dose. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel E: MK-7602 Single dose Part 1 (Experimental): Participants are inoculated with P. falciparum. Panel E participants receive MK-7602 as a single oral dose. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel F: MK-7602 Multiple dose Part 2 (Experimental): Participants are inoculated with P. falciparum. Panel F participants receive MK-7602 at multiple oral doses. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel G: MK-7602 Multiple dose Part 2 (Experimental): Participants are inoculated with P. falciparum. Panel G participants receive MK-7602 at multiple oral doses. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil
- Panel H: MK-7602 Multiple dose Part 2 (Experimental): Participants are inoculated with P. falciparum. Panel H participants receive MK-7602 at multiple oral doses. Participants will receive artemether/lumefantrine oral tablets as definitive antimalarial treatment. Additional definitive antimalarial treatment may be administered at the investigator's discretion.
  Interventions: Other: Plasmodium falciparum; Drug: MK-7602; Drug: Artemether/lumefantrine; Drug: Primaquine; Drug: Artesunate; Drug: Atovaquone/proguanil

INTERVENTIONS:
Other: Plasmodium falciparum — Parasite inoculation administered by intravenous (IV) infusion as the challenge agent
  Other Names: P. falciparum
Drug: MK-7602 — Capsules to be administered orally.
Drug: Artemether/lumefantrine — Tablets to be administered orally as definitive antimalarial treatment.
  Other Names: Riamet®; Coartem®
Drug: Primaquine — Tablets to be administered orally as definitive antimalarial treatment.
  Other Names: Primacin®
Drug: Artesunate — Intravenous (IV) infusion to be administered as definitive antimalarial treatment.
Drug: Atovaquone/proguanil — Tablets to be administered orally as definitive antimalarial treatment.
  Other Names: Malarone ®

SUMMARY:
The purpose of this study is to assess the antimalarial activity, pharmacokinetics, and safety of MK-7602 in healthy adults following Plasmodium falciparum (P. falciparum) infection.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Is in good health
* Has a body mass index (BMI) between 18 and 32 kg/m2, inclusive
* For participant assigned male sex at birth: If capable of producing sperm, participant must agree to the following during the study treatment period and for at least 90 days after the last dose of MK-7602: Refrain from donating sperm, plus EITHER be abstinent OR must agree to use male condom plus additional contraceptive method
* For participant assigned female sex at birth: EITHER be a person of nonchildbearing potential (PONCBP) OR must use a highly effective contraceptive method or be abstinent during the intervention period and for at least 10 days after the last dose of study intervention
* Must provide confirmation of not living alone (at any stage from inoculation day until the end of the study). A participant who lives alone may be included on a case-by-case basis.
* Agrees to refrain from eating food containing poppy seeds for 48 hours prior to screening, malaria inoculation, and MK-7602 administration

Exclusion Criteria:

* History of clinically significant clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated or has a history of clinically significant psychiatric disorder
* History of cancer (malignancy)
* History of malaria
* History of splenectomy
* History of ever receiving a blood transfusion
* History of recurrent headache (eg, tension-type, cluster or migraine) with a frequency of ≥2 episodes per month on average and severe enough to require medical therapy, during the 5 years preceding the screening visit
* History of convulsion (including intravenous drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood is not considered an exclusion criterion.
* Has presence of clinically significant infectious disease or fever (eg, sublingual temperature ≥38.5 degrees Celsius) within the 5 days prior to inoculation
* Has evidence of acute illness within the 4 weeks prior to screening that the Investigator deems may compromise participant safety
* Has clinically significant disease or any condition or disease that might affect drug absorption, distribution, or excretion (eg, gastrectomy, diarrhea)
* Has a medical requirement for intravenous immunoglobulin or blood transfusions
* Has had a major surgery with more than 470 mL of blood loss, lost 1 unit of blood (approximately 470 mL) or undergone blood donation of any volume to the Australian Red Cross Blood Service (Blood Service) or other blood blank within 4 weeks prior to the prestudy screening visit) or during the 8 weeks prior to inoculation
* Has used any corticosteroids, anti-inflammatory drugs (excluding commonly used over-the-counter anti-inflammatory drugs such as ibuprofen, acetylsalicylic acid, diclofenac), immunomodulators or anticoagulants within the past three months
* History of receiving immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone, or inhaled steroids) at a dose or duration potentially associated with hypothalamic-pituitary-adrenal axis suppression within the past year from the screening visit
* Has had any vaccination within the last 28 days
* Has participated in another investigational study within 12 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit
* History of participation in a previous malaria challenge study or malaria vaccine study.
* Must not have had malaria exposure that is considered by the principal investigator or their delegate to be significant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Parasite reduction ratio (PRR48) (Parts 1 and 2) | Pre-inoculation on Day 0, once daily Days 4 to 7, pre-dose of MK-7602 on Day 8, post-first dose of MK-7602 at 2, 4, 8, 12, 16, 24, 30, 36, 48, 54, 60, 72, (78 Part 2 only), 84, and 96 hours, and once daily Days 13, 15, 17, 20, 22, 24, 27, 29, 31, and 34
  PRR48 is the logarithm of the parasite reduction ratio per 48 hours determined from parasitemia data from time 0 to time 48 hours. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the PRR48.
Parasite Clearance Half-life (PCt1/2) (Parts 1 and 2) | Pre-inoculation on Day 0, once daily Days 4 to 7, pre-dose of MK-7602 on Day 8, post-first dose of MK-7602 at 2, 4, 8, 12, 16, 24, 30, 36, 48, 54, 60, 72, (78 Part 2 only), 84, and 96 hours, and once daily Days 13, 15, 17, 20, 22, 24, 27, 29, 31, and 34
  PCt1/2 is the half-life of the log-linear portion of the parasite clearance curve. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the PCt1/2.
Parasite Regrowth (Parts 1 and 2) | Pre-inoculation on Day 0, once daily Days 4 to 7, pre-dose of MK-7602 on Day 8, post-first dose of MK-7602 at 2, 4, 8, 12, 16, 24, 30, 36, 48, 54, 60, 72, (78 Part 2 only), 84, and 96 hours, and once daily Days 13, 15, 17, 20, 22, 24, 27, 29, 31, and 34
  Parasite regrowth is defined as initial parasite clearance followed by asexual parasite regrowth above 5,000 parasites/mL. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the parasite regrowth.
Part 1 Single dose: Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the AUC0-inf for Part 1.
Part 1 Single dose: Maximum Plasma Concentration (Cmax) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Cmax for Part 1.
Part 1 Single dose: Concentration at 24 Hours (C24) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the C24 for Part 1.
Part 1 Single dose: Time to Maximum Plasma Concentration (Tmax) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Tmax for Part 1.
Part 1 Single dose: Elimination Half-life (t1/2) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the t1/2 for Part 1.
Part 2 Multiple dose: Area Under the Curve Time 0 to End of the Dosing Interval (AUC0-tau) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-first dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72, 78, 84 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the AUC0-tau for Part 2.
Part 2 Multiple dose: Maximum Plasma Concentration (Cmax) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-first dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72, 78, 84 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Cmax for Part 2.
Part 2 Multiple dose: Time to Maximum Plasma Concentration (Tmax) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-first dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72, 78, 84 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Tmax for Part 2.
Part 2 Multiple dose: Elimination Half-life (t1/2) of MK-7602 | Pre-dose of MK-7602 on Day 8 and post-first dose of MK-7602 at 0.5, 1, 2, 3, 4, 8, 12, 24, 30, 36, 48, 54, 60, 72, 78, 84 and 96 hours and then once daily on Days 13, 15, 17, 20, and 22
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the t½ for Part 2.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to Day 45
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to Day 13
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- USC Clinical Trials Brisbane (South Bank) ( Site 0001), South Brisbane, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com